CLINICAL TRIAL: NCT06294600
Title: Biomarker-Guided Early Elarithromycin Treatment to Prevent Sepsis Progression in Community-Acquired Pneumonia: The React Randomized Clinical Trial
Brief Title: Clarithromycin Treatment to Prevent Sepsis Progression in CAP (REACT)
Acronym: REACT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REACT; 2023-507295-40 (EudraCT Number)
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Community-acquired Pneumonia
Keywords: CAP; CLARITHROMYCIN; SEPSIS; suPAR; PCT; ACCESS; SOFA; RSS
MeSH Terms: conditions — Community-Acquired Pneumonia; Sepsis | interventions — Clarithromycin; Tablets

STUDY DESIGN:
Intervention Model Description: This is a prospective, 1:1 randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): These patients will be treated with 1 placebo tablet every 12 hours and it is suggested that all patients receive at least one of antibiotics based on the current ESCMID guidelines for severe CAP13 (Ampicillin/sulbactam, Amoxicillin/clavulanate, Piperacillin/tazobactam, Ceftriaxone, Cefotaxime, Ceftaroline, Moxifloxacin). The total duration of treatment will be seven days.Τhe dosage, the dosage regime, the route and mode of administration, and the treatment period for the aforementioned antibiotics can be found in the relevant SmPCs (available in References). However, the attending physician may modify the antimicrobial treatment based on risk factors for multidrug-resistance pathogens, microbiology results and local epidemiology. All SoC treatment products and clarithromycin are authorised for use in Greece, where the trial will be conducted.
  Interventions: Drug: Tablets
- Clarithromycin (Active Comparator): These patients will be treated with oral clarithromycin 500 mg twice daily for seven days and it is suggested that all patients receive at least one of antibiotics based on the current ESCMID guidelines for severe CAP13 (Ampicillin/sulbactam, Amoxicillin/clavulanate, Piperacillin/tazobactam, Ceftriaxone, Cefotaxime, Ceftaroline, Moxifloxacin). The total duration of treatment will be seven days.Τhe dosage, the dosage regime, the route and mode of administration, and the treatment period for the aforementioned antibiotics can be found in the relevant SmPCs (available in References). However, the attending physician may modify the antimicrobial treatment based on risk factors for multidrug-resistance pathogens, microbiology results and local epidemiology. All SoC treatment products and clarithromycin are authorised for use in Greece, where the trial will be conducted.
  Interventions: Drug: Clarithromycin 500mg

INTERVENTIONS:
Drug: Clarithromycin 500mg — Oral tablets of 500mg of clarithromycin
  Other Names: A β-lactam/β-lactamase inhibitor or a 3rd generation cephalosporin or a fluoroquinolone
  Arms: Clarithromycin
Drug: Tablets — Oral tablets of similar appearance to active study drug
  Other Names: A β-lactam/β-lactamase inhibitor or a 3rd generation cephalosporin or a fluoroquinolone
  Arms: Placebo

SUMMARY:
The primary objective of the REACT randomized clinical trial (RCT) is to optimize the clinical benefit from adjunctive clarithromycin treatment shown in the ACCESS trial and to provide evidence for the clinical benefit of early start of adjunctive oral clarithromycin guided by suPAR to prevent the progression into sepsis in patients with community-acquired pneumonia (CAP) at risk. This can be achieved by endpoints incorporating clinical benefit with the effect of treatment on the improvement of the immune dysregulation of CAP. The secondary objectives of REACT are to investigate the impact of early adjunctive treatment with clarithromycin on the resolution of CAP at the test-of-cure (TOC) visit.

DETAILED DESCRIPTION:
Sepsis is recognized nowadays as one of the major causes of global morbidity and mortality. One analysis of global data revealed that 49 million of new cases are admitted to hospitals every year and that 11 million of the patients die. Sepsis is the life-threatening organ dysfunction which develops due to the dysregulated response of the host to an infection; mortality is ranging between 20 and 25%. The most common infections leading to sepsis are infections of the lower respiratory tract (LRTIs) mainly community-acquired pneumonia (CAP).

Numerous attempts have been done the last decades to decrease the substantial mortality of sepsis. Standard-of-care (SoC) therapy for sepsis is framed by the Surviving Sepsis Campaign (SSC) guidelines which are published every four years since 2004 (last publication 2021). The backbone of these guidelines is the early administration of intravenous antibiotics and fluids. In all editions of the SSC guidelines "early" means less than one hour from sepsis recognition. The experts recognize that the secret to decrease mortality is to intervene early before the dysregulated host response to the infection becomes exaggerated and impossible to withhold. The experts state that for every hour of delay in intervention the odds for survival decrease by relative 7.6%. Then the real ambiguity moves on how the initiation of the sepsis process can be recognized earlier than clinical deterioration appears.

The only way to achieve our current strategy is to implement a strategy linking the increase of a biomarker to an early intervention. This biomarker can be either a measured circulating protein or a bioscore. An example of how this strategy works is the biomarker-guided treatment of early COVID-19 (coronavirus disease 2019) recently approved by the European Medicines Agency (EMA). The biomarker suPAR (soluble urokinase plasminogen activator receptor) was used as a tool to recognize the patient at risk for severe respiratory failure and guided the start of the drug anakinra. This led to an overall 64% clinical benefit so as to become the first early precision intervention approved for infections by the EMA. The registered cut-off of suPAR which guides early intervention is 6 ng/ml or more.

The suPAR assay is not commercially available in the United States. However, all enrolled patients in SAVE-MORE trial were required to have a plasma soluble urokinase plasminogen activator receptor (suPAR) level ≥ 6 ng/mL. SAVE-MORE was double-blind, randomized controlled trial evaluated the efficacy and safety of anakinra, an IL-1α/β inhibitor, in 594 patients with COVID-19 at risk of progressing to respiratory failure as identified by plasma suPAR ≥6 ng ml-1, 85.9% (n = 510) of whom were receiving dexamethasone. In order to identify a comparable population as was studied in the SAVE-MORE trial, an alternative patient identification method was developed by the Food and Drug Administration (FDA) of the United States to select patients most likely to have suPAR ≥ 6 ng/mL based on commonly measured patient characteristics (Appendix I). This score contains eight clinical variable and patients meeting at least 3 of the variables should receive early anakinra treatment. Patients meeting at least three of the following eight criteria are considered likely to have suPAR ≥ 6 ng/mL at baseline: i) age 75 years or more; ii) need for oxygen supplementation; iii) current/previous smoking status; iv) Sequential Organ Failure Assessment (SOFA) score 3 or more; v) neutrophil-to-lymphocyte ratio (NLR) 7 or more; vi) blood hemoglobin 10.5 g/dL or less; vii) medical history of ischemic stroke; and viii) blood urea 50 mg/dL or more and/or medical history of renal disease. According to the SmPC, suPAR is a biomarker is used at the Emergency Department (ED) for the triage of patients for early discharge home or not; levels exceeding 6ng/ml advise for hosptialization.

With this precision-embedded approach adjunctive treatments may attenuate the exaggerated response of the host and improve outcomes. Macrolides are a unique class of drugs that combine both antibiotic and anti-inflammatory properties. Several meta-analyses have proven that addition of a macrolide to treatment decreases mortality by community-acquired pneumonia (CAP). However, the mortality benefit from macrolides treatment is coming from meta-analyses and no randomized clinical trial (RCT) has been published so far to demonstrate such a benefit. This is also heavily criticized in the recently published guidelines by the European Society of Intensive Care with the European Society of Clinical Microbiology and Infections Diseases (ESCMID) for the management of severe CAP where the recommendation for the co-administration of macrolides to β-lactams is characterized as low-quality evidence.

The only available RCT testing the value of early intervention with macrolides in patients with community-acquired pneumonia (CAP) is ACCESS (A randomized clinical trial of oral Clarithromycin in Community-acquired pneumonia to attenuatE inflammatory responseS and improve outcomeS) (EudraCT number 2020-004452-15; ClinicalTrials.gov NCT04724044). The inclusion criteria of the ACCESS trial have the characteristics of precision therapy i.e. participants were adults with CAP, meeting at least two of the criteria of the systemic inflammatory response syndrome, with SOFA (sequential organ failure assessment) score 2 or more and circulating procalcitonin 0.25 ng/ml or more. ACCESS had a composite primary endpoint pointing towards an early anti-inflammatory clinical benefit of clarithromycin. Patients achieving the endpoint should meet both two conditions A and B by day 4 since start of the study drug: condition A defined as at least 50% decrease of the respiratory symptoms score (RSS); and condition B defined as at least 30% decrease of the baseline SOFA score and/or favorable PCT kinetics (defined as at least 80% decrease of the baseline PCT or PCT less than 0.25 ng/ml). The study succeeded in the primary endpoint since this was met in 38.3% of patients randomized to the SoC + placebo group and in 67.9% of patients randomized to the SoC + clarithromycin group (p<0.0001). The ACCESS study also showed remarkable efficacy in all secondary endpoints and mainly to those endpoints pointing towards prevention of sepsis progression:

11.30% of patients treated with SoC and placebo progressed into sepsis during the 28-day follow-up compared to only 2.25% of patients treated with oral clarithromycin and placebo (hazard ratio 0.19; p: 0.009) 27.8% of patients treated with SoC and placebo developed a new sepsis episode during the 28-day follow-up compared to only 14.8% of patients treated with oral clarithromycin and placebo (hazard ratio 0.48; p: 0.009); and 65.4% of patients treated with SoC and placebo were discharged from hospital alive compared to 78.4% of patients treated with oral clarithromycin and placebo (hazard ratio 1.38; p: 0.027) Post-hoc analysis showed that 87.4% of study participants were meeting at least 3 of the FDA clinical score making the participants at high likelihood for suPAR 6 ng/ml or more. This means that use of suPAR can discriminate early patients with CAP who are at high likelihood to receive benefit towards prevention of progression into sepsis and organ dysfunction through early start of clarithromycin treatment.

Data from the ACCESS study also showed a significant effect of clarithromycin treatment on modulation of immune dysregulation taking place in CAP by day 4 when the primary endpoint was met. These data points towards improvement of the function of circulating monocytes towards better production of TNFα (tumour necrosis factor-alpha) after stimulation, decrease of circulating interleukin (IL)-10 and improvement of the IL-8/IL-10 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or above 18 years
* Male or female gender
* In case of women of reproductive age, willingness to use dual contraceptive method during the study period
* Written informed consent provided by the patient. For subjects without decision-making capacity, informed consent must be obtained from a legally designated representative following the national legislation
* Community-acquired pneumonia (CAP)
* Presence of at least two of the following signs: i) cough; ii) purulent sputum expectoration; iii) dyspnea; and/or iv) pleuritic chest pain
* PCT ≥0.25 ng/ml
* suPAR ≥6 ng/ml

Exclusion Criteria:

* Age below 18 years
* Denial of written informed consent
* Any stage IV malignancy
* Any do not resuscitate decision
* Patients necessitating non-invasive ventilation or mechanical ventilation
* Hospitalization in Intensive Care Unit
* Infection by SARS-CoV-2
* Oral or IV intake of corticosteroids at a daily dose equal to or greater than 0.4 mg/kg prednisone for a period greater than the last 15 days
* Intake of any macrolide for the current episode of CAP under study
* Known infection by the human immunodeficiency virus
* Any chronic anti-cytokine treatment for more than two months
* QTc interval at rest in the ECG ≥500 msec or history of know long QT syndrome
* Medical history of allergy to macrolides
* Concomitant oral intake of astemizole, cizapride, doperidone, pimozide, terfenadine, midazolam, ranolazine, ergot alkaloids (e.g. ergotamine and dihydroergotamine), lomitapide and colchicine; patients may be enrolled in the trial if they stop these drugs during trial participation.
* Medical history of torsades de pointes arrhythmia
* Concomitant intake of lovostatin or simvastatin; patients may be enrolled in the trial if they stop these drugs during trial participation.
* Concomitant presence of end-stage liver failure and end-stage renal failure.
* Severe hypokalemia or severe hypomagnesemia; a patient may be enrolled one any of these electrolyte disturbances are restored.
* Any contradictions for macrolide uptake
* Pregnancy or lactation. Women of child-bearing potential will be screened by a urine pregnancy test before inclusion in the study
* Participation in any other interventional trial within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-04-05 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Change of baseline respiratory symptoms score | 4 Days
  At least 50 percent (%) decrease of the sum of scoring (0-12) for the symptoms of cough (0-3), dyspnea (0-3), purulent sputum expectoration (0-3) and pleuritic chest pain (0-3) between baseline and Study Day 4
Change of baseline total sequential organ failure assessment (SOFA) score | 4 Days
  At least 30 percent (%) decrease between baseline sequential organ failure assessment (SOFA) score and measured sequential organ failure assessment (SOFA) score at Study Day 4.
Change of baseline on both plasma PCT and plasma IL-10 or IL-8 to IL-10 ratio | 4 Days
  Plasma PCT on visit 4 has decreased by at least 80% from baseline PCT on screening or it is below 0.25 ng/ml AND ([plasma IL-10 on visit 4 has decreased by at least 25% from IL-10 of visit 1 or it is below the lower limit of detection] OR [the IL-8 to IL-10 ratio of day 4 has decreased less than 15% from the IL-8 to IL-10 ratio of visit 1]).

SECONDARY OUTCOMES:
The number of patients that succeeded the resolution of CAP at the test of cure (TOC) visit. | 14 Days
  This is also analyzed separately for patients infected or colonized by clarithromycin-susceptible and clarithromycin-resistant S.pneumoniae and it is defined as the complete resolution of RSS
Need for up-escalation of the SoC administered antibiotics. | 28 Days
  This is considered as the change of the baseline administered SoC antibiotics into more broad-spectrum antibiotics.
Survival | 28 Days
  Alive hospital discharge until day 28
Change of baseline sequential organ failure assessment (SOFA) score | 8 Days
  Achievement of more than 50% decrease of baseline SOFA score at end-of-treatment (EOT) visit
Change of baseline on both plasma PCT and plasma IL-10 or IL-8 to IL-10 ratio | 8 Days
  Score of improvement of CAP-associated immune dysregulation (see sections of Laboratory procedures) at the end-of-treatment (EOT) visit
Cytokine production | 4 Days
  Change of cytokine production by PBMCs on day 4 from visit 1
28-Day Mortality | 28 Days
  Association of 28-day mortality with the score of improvement of CAP-associated immune dysregulation
90-Day Mortality | 90 Days
  Association of 90-day mortality with score of improvement of CAP-associated immune dysregulation
Cost | 90 Days
  Cost of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos J Giamarellos-Bourboulis, MD, Phd, Study Chair — Hellenic Sepsis Study Group
Locations (24):
- Greece (24):
  - 5th Pulmonary Department, SOTIRIA Athens General Hospital of Chest Diseases, Athens, Athens
  - 1st Department of Internal Medicine - General Hospital of Athens "Sismanogleio-Amalia Fleming", Athens, Greece
  - 1st Department of Internal Medicine, AHEPA University General Hospital of Thessaloniki, Athens, Greece
  - 1st Department of Internal Medicine, EVANGELISMOS Athens General Hospital, Athens, Greece
  - 1st Department of Internal Medicine, G. GENNIMATAS Athens General Hospital, Athens, Greece
  - 1st Department of Internal Medicine, General University Hospital of Ioannina, Athens, Greece
  - 1st Department of Internal Medicine, KORGIALENEIO-BENAKEIO E.E.S. Athens General Hospital, Athens, Greece
  - 1st Department of Internal Medicine, THRIASIO General Hospital of Elefsis, Athens, Greece
  - 1st University Department of Pulmonary Medicine, SOTIRIA General Hospital of Chest Diseases of Athens, Athens, Greece
  - 2nd Department of Internal Medicine, Attikon University Hospital, Athens, Greece
  - 2nd Department of Internal Medicine, THRIASIO General Hospital of Elefsis, Athens, Greece
  - 2nd Department of Internal Medicine, TZANEIO Piraeus General Hospital, Athens, Greece
  - 2nd Department of Internal Medicine, University General Hospital of Alexandroupolis, Athens, Greece
  - 3rd Department of Internal Medicine - General State Hospital of Nikaia "Saint Panteleimon" - West Attica General Hospital, Athens, Greece
  - 3rd Department of Internal Medicine, General Hospital of Athens KORGIALENEIO- BENAKEIO E.E.S., Athens, Greece
  - 3rd University Department of Internal Medicine, SOTIRIA Athens General Hospital of Chest Diseases, Athens, Greece
  - 4th Department of Internal Medicine, Attikon University Hospital, Athens, Greece
  - 6th Pulmonary Medicine Department, SOTIRIA General Hospital of Chest Diseases of Athens, Athens, Greece
  - Department of Chest Medicine, EVANGELISMOS Athens General Hospital, Athens, Greece
  - Department of Internal Medicine, Larissa University General Hospital, Athens, Greece
  - Department of Internal Medicine, Patras University General Hospital, Athens, Greece
  - Department of Pulmonary Medicine, General Hospital of Kerkira, Athens, Greece
  - Emergency Department, TZANEIO Piraeus General Hospital, Athens, Greece
  - 3rd Department of Internal Medicine, PAPAGEORGIOU General Hospital of Thessaloniki, Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: No